CLINICAL TRIAL: NCT00754884
Title: Phase IV Study of Nasal Salmon Calcitonin in the Treatment of Symptoms and Signs of Fibromyalgia
Brief Title: Calcitonin in the Treatment of Fibromyalgia
Acronym: CALFI
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Study drug was not longer available in our country.
Sponsor: Unidad de Investigacion en Enfermedades Cronico-Degenerativas (Other)
Responsible Party: Principal Investigator, Cesar Ramos Remus, M.D, Director, Unidad de Investigacion en Enfermedades Cronico-Degenerativas
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: UIECD-010
Record Dates: First submitted 2008-09-16; First posted 2008-09-18 (Estimated); Last update posted 2015-12-04 (Estimated); Status verified 2015-12

CONDITIONS: Fibromyalgia
Keywords: salmon calcitonin; endorphins; treatment; fibromyalgia
MeSH Terms: conditions — Fibromyalgia | interventions — salmon calcitonin; Glycerol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): 200 U.I. of intranasal salmon calcitonin
  Interventions: Drug: salmon calcitonin
- B (Placebo Comparator): intranasal saline solution and glycerol
  Interventions: Drug: intranasal saline solution plus glycerol

INTERVENTIONS:
Drug: salmon calcitonin — daily intranasal 200 U.I. salmon calcitonin for periods of 14 days at a time
  Other Names: Miacalcic nasal spray (Novartis Pharmaceutical)
  Arms: A
Drug: intranasal saline solution plus glycerol — daily intranasal (one shot) saline solution plus glycerol for a period of 14 days
  Other Names: Nasalub
  Arms: B

SUMMARY:
The purpose of this study is to determine whether nasal administration of salmon calcitonin is effective and safe in the treatment of symptoms and signs of primary fibromyalgia.

DETAILED DESCRIPTION:
Fibromyalgia is a common, chronic musculoskeletal disorder that is characterized by widespread pain and tenderness. Fibromyalgia occurs in around 2% of the US general population, is more common in women and is associated with substantial morbidity and disability. Treatment of fibromyalgia has been disappointing; roughly one-third of patients have had a clinically important therapeutic response to medications or no-medicinal treatment, event with the newest drugs reported in the literature. Pathophysiology of fibromyalgia is unknown, but abnormalities in central neurotransmission might play a role. Some studies have shown that salmon calcitonin increases peripheral and central levels of endorphins. Increasing endorphins levels may decrease pain. Then, it is feasible that nasal administered salmon calcitonin may decrease several of the symptoms and signs of patients suffering fibromyalgia.

ELIGIBILITY:
Inclusion Criteria:

* Female patients between 18 and 50 years
* Fibromyalgia diagnosis (ACR criteria)
* Must be able to apply the nasal medication
* Must be able to comply with study visits
* Must be able to understand informed consent
* Must be able to answer self-administered questionnaires
* Must have an active disease(VAS > 60mm)

Exclusion Criteria:

* Comorbid conditions (i.e. hypothyroidism, diabetes mellitus, etc.)
* Any disturbance in the nasal tissue
* Use of concomitant opioid analgesics
* Contraindication to use salmon calcitonin (allergy, hypocalcemia, hypophosphatemia)
* Other rheumatic diseases
* Diagnosis of major depressive disorder

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2008-10; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Functional status as assessed by the Fibromyalgia Impact Questionnaire (FIQ), a self-report inventory developed to measure health status in patients with fibromyalgia | Day 0, Day 14, Day 28 and Day 56

SECONDARY OUTCOMES:
Health related quality of life as assessed by WHO-DAS II, self-report questionnaire. Dolorimetry will be also used | Day 0, Day 14, Day 28 and Day 56

CONTACTS AND LOCATIONS:
Overall Officials: Cesar R. Ramos-Remus, M.D., MSc, Principal Investigator — Attending Rheumatologist HGR45 and Director UIECD
Locations (1):
- Hospital General Regional No. 45, IMSS, Guadalajara, Jalisco, Mexico

REFERENCES:
- [Background] Burckhardt CS, Clark SR, Bennett RM. The fibromyalgia impact questionnaire: development and validation. J Rheumatol. 1991 May;18(5):728-33. PMID 1865419
- [Background] Wolfe F, Smythe HA, Yunus MB, Bennett RM, Bombardier C, Goldenberg DL, Tugwell P, Campbell SM, Abeles M, Clark P, et al. The American College of Rheumatology 1990 Criteria for the Classification of Fibromyalgia. Report of the Multicenter Criteria Committee. Arthritis Rheum. 1990 Feb;33(2):160-72. doi: 10.1002/art.1780330203. PMID 2306288
- [Background] MacIntyre I, Alevizaki M, Bevis PJ, Zaidi M. Calcitonin and the peptides from the calcitonin gene. Clin Orthop Relat Res. 1987 Apr;(217):45-55. PMID 3549095
- [Background] Szanto J, Jozsef S, Rado J, Juhos E, Hindy I, Eckhardt S. Pain killing with calcitonin in patients with malignant tumours. Oncology. 1986;43(2):69-72. doi: 10.1159/000226336. PMID 3513074
- [Background] Mystakidou K, Befon S, Hondros K, Kouskouni E, Vlahos L. Continuous subcutaneous administration of high-dose salmon calcitonin in bone metastasis: pain control and beta-endorphin plasma levels. J Pain Symptom Manage. 1999 Nov;18(5):323-30. doi: 10.1016/s0885-3924(99)00081-0. PMID 10584455
- [Background] Gennari C. Analgesic effect of calcitonin in osteoporosis. Bone. 2002 May;30(5 Suppl):67S-70S. doi: 10.1016/s8756-3282(02)00713-5. PMID 12008161
- [Background] Ofluoglu D, Akyuz G, Unay O, Kayhan O. The effect of calcitonin on beta-endorphin levels in postmenopausal osteoporotic patients with back pain. Clin Rheumatol. 2007 Jan;26(1):44-9. doi: 10.1007/s10067-006-0228-z. Epub 2006 Mar 31. PMID 16575494
- [Background] Wolfe F. The fibromyalgia syndrome: a consensus report on fibromyalgia and disability. J Rheumatol. 1996 Mar;23(3):534-9. No abstract available. PMID 8832998
- [Background] Bessette L, Carette S, Fossel AH, Lew RA. A placebo controlled crossover trial of subcutaneous salmon calcitonin in the treatment of patients with fibromyalgia. Scand J Rheumatol. 1998;27(2):112-6. doi: 10.1080/030097498440976. PMID 9572636